CLINICAL TRIAL: NCT00789412
Title: SSI for Monitoring of Analgesia and Sedation in Critically Ill Patients
Brief Title: Surgical Stress Index as a Tool for Monitoring Analgesia and/or Sedation in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Berthold Bein, UKSH, Campus Kiel
Other Study IDs: SSI-154-01
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Analgesia; Sedation; Mechanical Ventilation; Pain; Stress; Intensive Care Unit; Critical Care
Keywords: Analgesia; Sedation; Critical Illness; Intensive Care
MeSH Terms: conditions — Agnosia; Pain; Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Expected ICU: Patients with expected postoperative admission to the ICU. Baseline measurement of SSI. Exploration prior to weaning.
- Unexpected ICU: Patients with unexpected stay at the ICU. No baseline measurement of SSI. Exploration in 'steady state' of analgosedation.

SUMMARY:
The hypothesis of the study is: Does the Surgical Stress Index (SSI) correlate with the Behavioral Pain Scale (BPS), the Ramsay Sedation Scale (RSS)and/or the Behavioral Pain Scale(BPV) and can therefore be used to monitor the quality of analgosedation in noncommunicative intensive care unit patients?

DETAILED DESCRIPTION:
The Surgical Stress index (SSI) was developed as a bedside tool to measure 'pain' during surgery. First trials showed a good correlation between SSI and aching procedures and a negative correlation to the dosage of Remifentanil. The first evaluation studies were performed under Propofol and Remifentanil anaesthesia. A different site of use for the Surgical Stress Index could be the intensive care medicine. 'Analgesia and Sedation are essential elements of intensive care treatment and relevant for patient outcome... There is therefore a need to monitor and define the level of sedation and pain and to provide the critically ill patient with adequate analgesia and sedation.' (j. martin 2002). Although the Ramsey Sedation Scale was never proven for validity and reliability it is an often used score for measurement of sedation quality. (Ramsay 74, Hansen-Flaschen 94, Jacobi 02, Martin 04). The Behavioral Pain Scale showed , apart from systolic blood pressure and heart rate, to be reliable and valid for measuring pain in noncommunicative, mechanical ventilated intensive care unit patients. (Payen 01, Jacobi 02, Aissaoui 05) These scales need to be performed a few times a day to be up to date and therefore time consuming for the intensive care staff. The Surgical Stress Index could be a non-invasive, bedside and online tool for measurement of sedation and/or analgesia in this complex patient group.

ELIGIBILITY:
Inclusion Criteria:

* analgosedated, mechanically ventilated patients on the ICU

Exclusion Criteria:

* neurological disorder
* age under 18
* lack of sinus rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: postoperative patients with admission to the intensive care unit who are intubated and mechanically ventilated
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Scholz, Prof Dr med, Study Chair — Institut für Anästhesiologie und Operative Intensivmedizin, Universitätsklinik Schleswig-Holstein, Campus Kiel
Locations (1):
- Institut für Anästhesiologie und Operative Intensivmedizin, Universitätsklinik Schleswig-Holstein, Campus Kiel, Kiel, Germany